## A CASE SERIES ON INCIDENTALLY DETECTED GALL BLADDER MALIGNANCY

Dr. Sathaiah Dadi\*, Dr. Meghana Maria Tharakan^, Dr. Perugu Venkateshwar\*, Dr. Swarajya^, Dr. Rithika TN\*,

Official Title of the Study: A CASE SERIES ON INCIDENTALLY DETECTED GALL BLADDER MALIGNANCY (Retrospective Analysis)

**NCT** number:

Date of the document: 08-08-2022

**Study period:** 01-01-2019 to 31-12-2019

## STUDY DESIGN, MATERIAL, AND METHODS:

A retrospective analysis of hospital records of patients who underwent Cholecystectomy in year duration (2019) for benign conditions, diagnosed and confirmed histopathologically as Gallbladder Malignancy. There are a total of one hundred and eighty patients who underwent cholecystectomy at our hospital (Osmania General Hospital) in 2019; out of which seven patient's histopathological diagnosis was gall bladder malignancy. We reviewed all the case's history and cross-checked the histopathological slides and confirmed the diagnosis. To avoid the bias of covid-19 pandemic in surgical practice we confined the patient records to the pre-pandemic period of one-year duration (2019).

**Case Series**: All the case details including the investigations and the final diagnosis are incorporated in the table format (Table-1)

Table- 1: Showing the details of patients diagnosed with gallbladder malignancy, and the final histopathological diagnosis

| Case<br>No | Gender | Age | Clinical presentation | Investigations | Procedure done | Histopathol ogy |
|---|---|---|---|---|---|---|
| 1 | Female | 60 | Right upper abdominal<br>pain, yellowish<br>discolouration of eyes,<br>Nausea for 10days | USG – Multiple calculi<br>with max diameter<br>6mm<br>CT – Cholelithiasis,<br>CBD diameter- 11mm | ERCP stenting Laparoscopic Cholecystectomy | Intestinal type<br>metaplastic<br>gallbladder<br>malignancy |
| 2 | Male | 65 | Right upper abdominal pain – 20days | USG – Distended<br>gallbladder with no<br>mass lesions and a<br>hypoechoic density | Open<br>Cholecystectomy | Adenocarcino ma gallbladder infiltrating muscularis mucosa |
| 3 | Female | 58 | Right upper abdominal pain radiating to back – 3 days | USG – Multiple calculi<br>and a small <1cm<br>polyp in the<br>gallbladder<br>CECT: 1*0.7cm polyp | Laparoscopic to<br>Open<br>cholecystectomy | Welldifferenti<br>ated<br>adenocarcino<br>ma of gall<br>bladder |
| 4 | Female | 40 | Right upper abdominal pain- 20 days | USG – 8*10mm polyp | Laparoscopic<br>Cholecystectomy | Welldifferenti<br>ated<br>adenocarcino<br>ma of gall<br>bladder |
| 5 | Male | 59 | Right upper abdominal pain- 20 days Lump in the upper abdomen- 20 days | USG – Distended<br>gallbladder with<br>Sludge<br>CECT – Thickened<br>gallbladder wall with<br>periGB collection S/O<br>Perforation | Open Subtotal<br>Cholecystectomy | Well to<br>moderately<br>differentiated<br>adenocarcino<br>ma of gall<br>bladder |
| 6 | female | 52 | Right upper abdominal pain- 20 days | USG- Distended gallbladder with no mass lesions | Laparoscopic to<br>Open<br>cholecystectomy | Welldifferenti<br>ated<br>adenocarcino<br>ma of gall<br>bladder |
| 7 | female | 55 | Right upper abdominal pain- 20 days | USG – Multiple calculi<br>with max diameter<br>6mm | Laparoscopic<br>Cholecystectomy | Welldifferenti<br>ated<br>adenocarcino<br>ma of gall<br>bladder |

## **Statistical Analysis:**

A total of 180 patients underwent cholecystectomy for various benign conditions in one year, out of which seven patients confirmed histopathologically with Gallbladder malignancy.

| Total no of | 180 |
|----------------|------|
| patients | |
| Diagnosed with | 7 |
| malignancy | |
| percentage | 3.8% |

Among these seven, three patients converted from laparoscopic to open procedure for difficulty with resection, two patients are posted for surgery considering empyema of gall bladder preoperatively, one patient posted in view of gall bladder perforation, and two patients preoperative diagnosis was gall bladder polyp.

| Converted from Lap to Open | 3 |
|----------------------------|---|
| Pre-op GB Polyp | 2 |
| Perforated GB | 1 |
| Empyema GB | 2 |

Only one patient is 40 years old and others are more than 50 years, and two of them are males.

| Total | 7 | Percentage |
|---------|---|------------|
| Males | 2 | 28.5 |
| Females | 5 | 71.5 |

Out of a total of 180 patients who underwent cholecystectomy, 117 are females and 63 are males

| Total | 180 |
|---------|-----|
| Males | 63 |
| Females | 117 |

Out of 180, the age distribution is as follows Percentage of malignancy detected

| Age | Percentage |
|---------|------------|
| 20 - 29 | 0 |
| 30 – 39 | 0 |
| 40 – 49 | 0.005 |
| >50 | 99.99 |

It implies that the malignancy rate increases with an increase in the patient's age more than 50 years and also with gender (Females > males)